CLINICAL TRIAL: NCT00546013
Title: Abdominal Aortic Aneurysms Are Associated With Pseudoexfoliation Syndrome
Brief Title: Abdominal Aortic Aneurysms and Pseudoexfoliation Syndrome
Status: Terminated | Type: Observational
Why Stopped: all patients required included
Sponsor: European Georges Pompidou Hospital (Other)
Other Study IDs: 01
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Abdominal Aortic Aneurysms; Pseudoexfoliation Syndrome; Hypertension
Keywords: abdominal aortic aneurysms; pseudoexfoliation syndrome; glaucoma
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Exfoliation Syndrome; Hypertension; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AAA group, control group: AAA group : with AAA Control group: without AAA

SUMMARY:
Conflicting results have been reported concerning the association of pseudoexfoliation syndrome (PXF) and abdominal aortic aneurysms (AAA). Schumacher et al. reported an association between AAA and PXF, with no consideration of grade. However, a later study did not confirm the association between AAA and PXF. The present study aimed at comparing the relative prevalence of PXF in patients suffering from AAA and in age-matched hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Presence of abdominal aortic aneurism
* Systemic hypertension without abdominal aortic aneurism over 60 years old

Exclusion Criteria:

* Unknown status for abdominal aortic aneurism

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in patients suffering from abdominal aortic aneurism as part of a routine clinical yearly follow-up and hypertensive patients without abdominal aortic aneurism and that were more than 60 years old to have similar mean ages in both groups, as pseudoexfoliation and abdominal aortic aneurism are age-related disorders
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2001-12; Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
standard ophthalmologic examination to group patients according to their pseudoexfoliation status | Day of standard ophthalmologic examination

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Rossignol, MD, PhD, Study Director
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France